CLINICAL TRIAL: NCT05779397
Title: Clinical Performance of Masimo Rad-GT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIP-1064
Record Dates: First submitted 2023-03-09; First posted 2023-03-22 (Actual); Results first posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-06

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Test Subject (Experimental): All subjects who are enrolled into the test group and participate in data collection receive the noninvasive Masimo RAD-GT
  Interventions: Device: Masimo RAD-GT

INTERVENTIONS:
Device: Masimo RAD-GT — Non-contact infrared thermometry device

SUMMARY:
The study is designed to validate the clinical performance of Masimo Rad-GT in the accuracy of temperature measurements.

DETAILED DESCRIPTION:
Individual sites are only representative of a subset of the overall population, per ISO 80601-2-56:2017(Medical electrical equipment - Part 2-56: Particular requirements for basic safety and essential performance of clinical thermometers for body temperature measurement), and therefore clinical bias and limits of agreement should not be evaluated for the subsets. Publication of results should include repeatability from individual sites and the combined clinical bias and limits of agreement (NCT05779397, NCT05787782, and NCT05674344).

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 to 80 years of age.
* Subjects are able to read and communicate in English as well as understand the study and the risks involved.

Exclusion Criteria:

* Subject is pregnant or nursing.
* Subject has a known neurological and/or psychiatric disorder (e.g., schizophrenia, bipolar disorder, Multiple Sclerosis, Huntington's disease) that interferes with the subject's level of consciousness. *
* Subject has any medical condition which in the judgment of the investigator and/or study staff, renders them ineligible for participation in this study or subject is deemed ineligible by the discretion of the investigator/study staff.

(* = Per study staff discretion)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Corporation, Irvine, California, United States

REFERENCES:
- See also: Validation of the Masimo INVSENSOR00063 in Febrile and Afebrile Subejcts — https://clinicaltrials.gov/ct2/show/NCT05787782?term=koei0004&draw=2&rank=1
- See also: Calibration and Validation of the Masimo Temperature Device in Febrile Patients — https://clinicaltrials.gov/ct2/show/NCT05674344?term=choc0008&draw=2&rank=1

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 68 enrolled participants, 68 completed the study.
Groups:
- Rad-GT: All subjects who are enrolled into the test group and participate in data collection receive the noninvasive Masimo RAD-GT
  Masimo RAD-GT: Non-contact infrared thermometry device
Period: Overall Study
Arm/Group | Rad-GT
Started | 68
Completed | 68
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Rad-GT
Number analyzed (Participants) | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 68
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 46
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Caucasian | 32
  Ethnicity: Hispanic | 5
  Ethnicity: Asian or Pacific Islander | 23
  Ethnicity: Other | 6
  Ethnicity: More than one | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 68

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Masimo Rad-GT Temperature Measurements (Degrees Celsius)
Description: The accuracy of the Masimo Rad-GT sensor will be determined by calculating the clinical bias (Δcb), limits of agreement (LA), and repeatability (σr). The temperature measurements from Masimo Rad-GT will be compared to the reference temperature measurements (Degrees Celsius).
Time Frame: 1-3 hours
Population: Data for 7 subjects was excluded as they did not complete at least one full one round of measurements.
  Data for 37 subjects was excluded as the data suggested existence of external conditions that interfere with RCT (reference clinical thermometer) or Rad-GT measurements.
Measure: Number; unit: Degrees Celsius
Arm/Group | Rad-GT
Number analyzed (Participants) | 24
Degrees Celsius
  Clinical Bias | -0.24
  Limits of Agreement | 0.85
  Repeatability | 0.04

ADVERSE EVENTS:
Time Frame: 1-3 hours
Arm/Group | Rad-GT
All-Cause Mortality (participants affected / at risk) | 0/68
Serious Adverse Events (participants affected / at risk) | 0/68
Other Adverse Events (participants affected / at risk) | 0/68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/97/NCT05779397/Prot_SAP_000.pdf